CLINICAL TRIAL: NCT07365124
Title: Developing and Optimising the Use of Magnetic Resonance Imaging and Spectroscopy in Radiotherapy (MRinRT) Pathways: Investigating Avenues to Improve Outcomes for Patients and the Assessment of Treatment Response.
Brief Title: MRinRT: Swansea University and SWWCC Collaboration Study.
Acronym: MRinRT
Status: Not yet recruiting | Type: Observational
Sponsor: Swansea Bay University Health Board (Other)
Collaborators: Swansea University (Other)
Responsible Party: Sponsor
Other Study IDs: SBU66
Record Dates: First submitted 2025-12-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma; Glioblastoma; Radiotherapy; MRI; MRI-guided Adaptive Radiotherapy; MRI Scanner Configuration; MRI Image Enhancement; Oesophageal Carcinoma; Pancreas Carcinoma; Gastric Cancer; Brain (Nervous System) Cancers
Keywords: MRI; Radiotherapy; MRI adaptive radiotherapy; MRI Imaging Biomarker
MeSH Terms: conditions — Carcinoma; Glioblastoma; Esophageal Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Neurologic Manifestations; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteer: Volunteers with no history of any medical issue which may affect the scan interpretation and who are eligible for MRI scanning
  Interventions: Other: MRI
- Patient: Patients with the tumour of interest who are due to undergo radiotherapy and are eligible for MRI scanning
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — This is an observational study with no interventions. Participants will undergo MRI scanning for research purposes and radiotherapy treatment will be delivered as per standard of care for the participants tumour type.

SUMMARY:
The aim of this study is to learn whether using MRI (magnetic resonance imaging) scans to plan radiotherapy is better than using CT (computed tomography) scans alone. The main questions it aims to answer is:

* Can MRI scan images be adjusted to make the tumour and normal tissues easier to see?
* Does adding MRI to a radiotherapy planning CT make the radiotherapy plan more precise?
* Can MRI be used to adjust a radiotherapy plan during a course of treatment to make it more precise, and might that reduce the side effects?
* Are there particular MRI scans that can predict how a tumour will respond to radiotherapy or how likely the patient is to have side effects?

This study will assess current MRI scanning procedures and ensure these are adjusted to best suit radiotherapy planning. It will also provide pilot data evaluating:

1. MRI-adapted radiotherapy Usually, radiotherapy plans are based on a pre-treatment planning CT scan. Unless an issue is detected the patient would complete their whole course of radiotherapy on this plan. This does not account for changes in position/size/shape of the tumour that occur over the whole treatment course. Clinicians therefore increase the size of the tumour/target to account for these uncertainties, which can increase side effects. This study will assess the potential to reduce side effects from radiotherapy by using repeat MRI scans and replanning during the treatment course (MRI-adaptive radiotherapy).
2. Imaging biomarkers MRI sequences can be used to predict response to radiotherapy or chance of developing side effects. This study will identify potential MRI sequences that may be used as imaging biomarkers, to guide the development of future clinical trials.

The study will be undertaken at SBUHB, lasting 4 years, and involving ≤15 healthy volunteers and ≤150 patients.

DETAILED DESCRIPTION:
Background Advances in radiotherapy technology have allowed treatments to become more conformal with steeper dose gradients, meaning target volumes are smaller and dose to surrounding normal tissues reduced. This is possible, in part, due to improvements in imaging used in radiotherapy planning and in the development of Intensity Modulated Radiotherapy. The current standard of care for most tumour sites is for target volumes to be delineated on a planning CT scan, with additional information from diagnostic imaging such as MRI or PET which can be fused with the planning CT scan. MRI is known to give clearer images of soft tissues and tissue planes allowing for more accurate target volume delivery. The fusion of MRI to the planning CT scan to aid target volume delineation is a standard of care for certain tumour sites, e.g. brain, but not in others such as oesophagogastric cancers.

Optimisation of MRI protocols for Novel Tumour sites Our group undertook a scoping review into the use of MRI for radiotherapy target volume delineation for gastric cancers and has found that although there is evidence of improved contrast resolution with MRI in comparison to CT, clinical utility for radiotherapy planning is yet to be demonstrated. The research group has also performed a pilot study assessing the addition MRI to CT planning scans for radiotherapy planning for gastric cancers which demonstrated potential for clinical benefit. The limitations of this study were small patient numbers and that MRIs used were diagnostic scans optimised for liver imaging rather than gastric cancers. An issue identified was poor anatomical correlation of the MRI to CT planning scan due to differences in stomach filling. Our study will build on this work to optimise the MRI sequences for improved clarity of imaging and to identify and standardise optimal pre-examination preparation.

It is possible to acquire a range of MRI sequences with each giving different information. Furthermore, contrast agents may be used during image acquisition to improve visualisation of the target of interest. The choice of contrast agent and sequences depends on whether the aim is to assess the size/location of the tumour or to assess a functional aspect of the tumour allowing the potential to act as a predictive or prognostic imaging biomarker. This study aims to optimise the choice of MRI sequences for target volume delineation in various anatomical regions and to assess the potential impact of MR imaging on radiotherapy planning in anatomical regions where it is not currently routine practice. In the UK there is an ongoing similar study that aims to optimise the MRI sequences for use on MRI-Linear Accelerator (MR-Linac) machines. Our study will follow similar principles in order to optimise MRI sequences for radiotherapy planning from stand-alone MRI scanners. The investigators postulate that our findings will be more generalisable compared to the recruiting MR-Linac study, as the vast majority of UK Oncology Centres do not have access to MR-Linac machines.

The potential for an MRI-Adaptive workflow Radical (curative-intent) or neoadjuvant radiotherapy treatment is often delivered as multiple treatment fractions given over several weeks. The current standard of care is to generate a radiotherapy plan based on a pre-treatment CT planning scan with guidance from additional diagnostic investigations depending on tumour site. Unless an issue is detected during treatment, e.g. detected by the on-treatment cone-beam CT(CBCT) set-up verification process, the patient would complete their whole course of treatment as per the radiotherapy plan based on the pre-treatment CT planning scan. This does not account for changes in the position, size or shape of the tumour that occur over the whole radiotherapy treatment course. Clinicians therefore add margins around the target volume to account for these potential uncertainties, leading to a larger target volumes and increased dose to surrounding normal structures, which can lead to increased toxicity. A potential solution to this issue could be to re-image and re-plan during the treatment course, termed 'adaptive radiotherapy'. MRI is already utilised for adapted radiotherapy workflow, particularly when an MR-Linac is available. This study will explore whether a diagnostic MRI may be used for RT plan adaptation. Of note, similar strategies have been assessed using CBCT with a 'plan of the day' approach in bladder cancer and there is also ongoing work assessing the benefit of adapting RT based on a mid-treatment PET scan in the PEARL study for oropharyngeal cancers.

Exploring Imaging Biomarkers MRI can also be used to determine quantitative information about functional biological processes, via the use of quantitative imaging biomarkers. These are defined as 'an objective characteristic derived from an in vivo image measured on a ratio or interval scale as an indicator of normal biological processes, pathogenic processes, or a response to a therapeutic intervention'. Current protocols include sequences which can be used to estimate functional characteristics of a tumour and surrounding tissues which could act as a biomarker to predict response to treatment or likelihood of a patient developing toxicity from treatment. However, there is limited validation of these biomarkers in clinical settings, in particular there is a lack of data assessing the repeatability and reproducibility.

Rationale and Risks/Benefits MRI is a non-invasive imaging technique which does not rely on ionising radiation exposure. It gives clearer images of soft tissues and tissue planes allowing for more accurate target volume delineation. More accurate delineation may allow clinicians to use smaller margins and therefore to spare surrounding normal tissues from radiotherapy induced damage thereby reducing toxicity.

This is a non-interventional, prospective study and therefore the investigators do not anticipate any serious adverse events directly relating to the scanning protocols. Standard MRI safety screening will be conducted to minimise the risk of serious adverse events such as those caused by permitting non-MR Safe individuals (as outlined in the exclusion criteria) to approach the magnetic field (e.g., malfunction of cardiac pacemaker). This study will investigate contrast enhanced sequences using licensed IV gadolinium-based contrast agents. These are widely used in clinical practice and are generally well tolerated but can present a risk of severe allergic reaction in 0.004%-0.7% patients and if given to patients with impaired renal function there is a risk of nephrogenic systemic fibrosis. Such contrast agents will be given to patients in line with the university's contrast agent policy and always under the supervision of a clinician.

Pre-examination participant preparation may be achieved through administration of oral contrast/filling agents. These can be used to improve visibility of the stomach lining and provide organ distention where appropriate. Most commonly, water has been administered but other food grade, non-medicinal contrast agents have been explored, most notably fruit juices e.g., pineapple and blueberry, or milk based drinks. Prior to administration, all participants will undergo an allergy check. Selecting the optimal oral contrast agent for MRI to aid radiotherapy planning will depend on factors such as disease location, purpose for which MRI sequences are to be obtained and importantly patient preference. There is currently limited published data regarding which is the optimal choice of oral contrast agent with respect to the imaging quality and also the patient experience of taking oral contrast agents for MRI scans.

For patients participating in this study, their radiotherapy planning will be as standard of care and their inclusion in the study not have any effect on their radiotherapy pathway.

Hypotheses

1. Optimisation of MRI protocols MRI protocols, including pre-examination participant preparation, may be optimised to support radiotherapy planning and applied to novel tumour sites and to tumour sites where MRI planning is already a standard of care.
2. Assess the effect of MRI-CT Integration in the radiotherapy pathway The integration of MRI with CT planning scans will enhance visualisation and accuracy of delineation of target volumes and organs at risk (OARs) and subsequent radiotherapy treatment planning, thereby enabling more precise treatment delivery and reducing radiotherapy-induced toxicity.
3. MRI-Adapted Radiotherapy MRI-adapted radiotherapy is feasible across multiple target sites and will improve clinical outcomes by enabling more accurate dose delivery, reducing radiation exposure to normal tissues, and consequently lowering treatment-related toxicity.
4. Imaging Biomarkers The investigators hypothesise current and novel MRI sequences are feasible, predictive and prognostic imaging biomarkers that can be developed and tested in the clinical setting. Quantitative MRI has the potential to assess of treatment response, inform clinical decision-making, and support patients in making more informed choices about their care.

Study Aims:

1. Optimisation of MRI protocols To have clinically-ready MRI protocols for use in clinical practice. This will entail optimising MRI sequences for radiotherapy planning, including optimising the pre-examination preparation and patient experience. Initial work will focus on 3 tumour sites

   1. Oesophago-gastric
   2. Pancreas
   3. Brain

   On completion of these subsites, proposed further anatomical sites include:
   * Head and Neck
   * Thorax - chest wall and breast
   * Thorax - lung
   * Abdomen
   * Pelvis - male
   * Pelvis - female
2. Assess the effect of MRI-CT Integration on quality of radiotherapy To determine if the addition of the information acquired from MRI, in addition to the current CT, will provide superior visualisation of the anatomy and extent of tumour, improving the accuracy of radiotherapy. The feasibility and clinical benefit of the addition of MRI will be determined by comparing the resulting delineation and subsequent dose distribution with that using CT alone.

Secondary Aims:

1. MRI-Adapted Radiotherapy To determine if repeat MRI scans undertaken during a course of radiotherapy can give additional information over CT alone, that will inform changes in the radiotherapy plan which lead to better outcomes for the patient. Radiotherapy plans at start and during treatment, using CT alone versus CT plus MRI scanning will be compared. The effect on dose distribution and the impact of this on tumour control and toxicity will be assessed.
2. Imaging Biomarkers Identify and develop structural and functional MRI sequences for use as imaging biomarkers in selected tumour sites. These biomarkers could be used to predict which patients may benefit from radiotherapy and/or assess the response to RT during and after treatment.

Study Design The study will consist of three parallel strands. These strands form the underpinning methodology for individual sub-studies which will investigate different tumour sites.

Strand 1 - Optimising MRI protocols and assessing the effect of MRI-CT integration in the radiotherapy pathway

This strand will progress over 4 stages:

1. Optimisation of MRI protocols: Healthy Volunteer Initial Imaging Studies of Normal Tissue Up to 15 healthy volunteers will be scanned to ascertain the best MRI sequences and parameters to obtain optimal images of the organ of interest. Pre-examination tissue preparation (e.g. stomach filling volumes and material) for abdominal MRI will also examined and optimised. Images will be assessed qualitatively for improvements in image quality, such as SNR and contrast. Trade-offs, such as increased examination time will also be considered to evaluate feasibility in a clinical setting. This stage will be considered complete once the success criteria below is achieved.
2. Optimisation of MRI protocols: Patient Volunteer Imaging Studies of Tumour/Normal Tissue Up to 20 patients per tumour site will be scanned alongside their standard treatment pathway to ascertain the best MRI sequences and parameters to obtain the highest quality images of the tumour and nearby organs of interest. Pre-examination tissue preparation (e.g. stomach filling volumes and material) for abdominal MRI will also examined and optimised. The goal would be to optimise images for improved expert rater acceptance and test feasibility of MRI for radiotherapy planning in patients. This stage will be considered complete once the success criteria is achieved.

   Predefined success criteria for each organ/tumour site for - Strand 1 stage a Healthy Volunteer and stage b Patient Volunteer Studies:
   1. - Participant acceptability The participant questionnaire responses will be reviewed to ensure acceptability. This is defined as an average score of 4 or higher on a 5-point Likert scale for MRI section Q1 and Q2 as shown in the Participant Questionnaire.
   2. - Two MRI physicists' opinions that sequences are adequately optimised to meet the requirements for radiotherapy planning.

      Assessment of sequences may include review of specific sequence parameters (following international guidance on MRI in RT) and geometric distortion characterisation. The MRI Characteristics will be recorded and the Physicist Team Questionnaire will be completed.
   3. - Visual grading characteristics analysis rating 4 or higher and deemed acceptable for clinical purposes The optimised sequences will then be reviewed by at least 3 independent expert clinicians in order to undertake visual characteristics grading analysis and determine if the images are clinically acceptable.
3. Assessing the effect of MRI-CT integration in the radiotherapy pathway: Tumour definition/Target Volume Delineation To assess the effect of MRI-CT Integration in the radiotherapy pathway, acquired MRI scans with be used alongside the patient's CT planning scan to determine the benefits of MRI in tumour delineation. This section of the study will evaluate target volume delineation with and without MRI to determine the clinical benefit of having MR images available and fused to the planning CT scan at the time of RT target volume delineation by assessing the changes in dosimetry and target volumes when RT is planned with vs without MRI. Conformity indices will be calculated to determine the level of agreement between the paired plans. The effects of including MRI on the confidence rating of the clinician outlining the target volumes will also be evaluated as per the Outlining Clinician Questionnaire.

   A minimum sample size of 10 patients with MRI scans will be acquired for these comparison studies.
4. Pathway Development Patients needing MRI for radiotherapy have particular requirements and this work aims to make MRI for radiotherapy as inclusive as possible. For example, the patients may not be able to tolerate long MRI scans and may not be able to tolerate breath-holds which are sometimes needed. They also may need to be immobilised in some way to ensure that they are being imaged in the same configuration that they will be imaged for their radiotherapy treatments. Qualitative surveys will be undertaken to assess patient acceptance of having an MRI as part of the radiotherapy treatment planning pathway as per the Participant Questionnaire in Appendix 6. Patient pathways will then be developed and integrated into standard clinical workflow for tumour sites where having MRI available at the time of RT planning has been shown to be beneficial.

Strand 2 - MRI-adapted radiotherapy Substudies will be developed in specific tumour sites to assess the utility of MRI during a course of radiotherapy (e.g. at the mid-point) to assess treatment response and allow for radiotherapy to be adapted for re-planning to focus on the residual tumour. The new plan will be compared to the original radiotherapy plan to determine the changes in target volume, dosimetry and dose to surrounding normal structures. Changes in predicted toxicity will be determined by using normal tissue complication models. If found to provide potential benefit in terms of predicted reduction in toxicity then this work would act as a pilot to guide the protocol of a future clinical trial to examine this further. A sample size of 10 patients will be acquired for these comparison studies.

Inclusion of patients in this study will be alongside their standard clinical pathway. Participating will not affect their standard radiotherapy pathway and the MRI obtained is purely for research purposes.

Strand 3 - Imaging biomarkers Sub-studies will evaluate MRI sequences that have the potential to act as functional biomarkers e.g. predicting response to treatment or likelihood of developing toxicity for selected tumour sites. For example, by using T2-weighted and DWI MRI sequences a measure of blood flow can be calculated and this is postulated to be predictive of response to radiotherapy.

Advanced sequences to be tested may include (but not confined to):

* Diffusion-weighted imaging (DWI) including "high-b value" imaging to assess tissue microstructure.
* Perfusion-weighted imaging and dynamic contrast enhanced imaging (DCE) to assess tumor microvasculature.
* Magnetic resonance spectroscopy (MRS) to assess the chemical biomarkers present in the tumour(s).

These images/spectra will then be analysed. Where feasible, the investigators will develop pilot studies that will compare to post-treatment outcomes, such as post-operative pathology, to assess the extent of tumour response to radiotherapy. This will allow identification of promising functional biomarkers which can then be studied in future research studies/clinical trials.

ELIGIBILITY:
Inclusion Criteria for health volunteers:

* Free from medical conditions that could confound imaging or study results
* Eligible for MRI

Inclusion Criteria for patients:

* Confirmed diagnosis of invasive carcinoma at the relevant tumour/target sites listed in this protocol
* Scheduled to receive radiotherapy to the target site
* ECOG performance status of 0-2
* Eligible for MRI (determined through MRI safety screening)

Exclusion Criteria:

* Presence of medical conditions that may interfere with study outcomes or data interpretation
* Use of regular medications that could affect imaging results or safety
* Any contraindications to MRI scanning, including but not limited to claustrophobia, reduced thermal regulatory capabilities, MR Unsafe implants and foreign bodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants for this study will be:
  1. healthy volunteers from Swansea Bay University Health Board or Swansea University
  2. patients with cancer who are due to undergo radiotherapy at Swansea Bay University Health Board
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Optimisation of MRI images 1 | From enrolment to analysis, on average 4-6 weeks
  Participant acceptability with average rating of 4 or higher on the Participant Questionnaire MRI Section Q1 and Q2
Optimisation of MRI images 2 | From enrolment to analysis, on average 4-6 weeks
  Physics team expert opinion that the sequence is optimised, assessed as per the Physics Team Questionnaire by 2 independent expert medical physicists
Optimisation of MRI images 3 | From enrolment to analysis, on average 4-6 weeks
  Visual grading characteristics analysis rating 4 or higher and deemed acceptable for clinical purposes by 3 independent clinicians as per the Image Properties Data Collection Form
Assess the effect of MRI-CT Integration in the radiotherapy pathway 1 | From enrolment to analysis, on average 4-6 weeks
  This will involve analysis of radiotherapy plans produced with and without an MRI scan at the time of the CT planning scan, to include:
  Dosimetry Comparison (evaluation of differences in dose distributions delivered to target volumes and OARs);
Assess the effect of MRI-CT Integration in the radiotherapy pathway 2 | From enrolment to analysis, on average 4-6 weeks
  This will involve analysis of radiotherapy plans produced with and without an MRI scan at the time of the CT planning scan, to include:
  Volumetric Comparison (assessment of differences in target and OAR delineation volumes);
Assess the effect of MRI-CT Integration in the radiotherapy pathway 3 | From enrolment to analysis, on average 4-6 weeks
  This will involve analysis of radiotherapy plans produced with and without an MRI scan at the time of the CT planning scan, to include:
  Qualitative Confidence Assessment (expert ratings of confidence in contouring accuracy rated on a 5-point Likert scale as per Outlining Clinician Questionnaire)
Assess the effect of MRI-CT Integration in the radiotherapy pathway 4 | From enrolment to analysis, on average 4-6 weeks
  This will involve analysis of radiotherapy plans produced with and without an MRI scan at the time of the CT planning scan, to include:
  Prediction of change in toxicity using normal tissue complication probability modelling

SECONDARY OUTCOMES:
MRI-Adapted Radiotherapy 1 | From enrolment to analysis, on average 4-6 weeks
  This will involve analysis of radiotherapy plans produced following an MRI scan during radiotherapy treatment and compared to the original radiotherapy plan, to include:
  Dosimetry Comparison (evaluation of differences in dose distributions delivered to target volumes and OARs);
MRI-Adapted Radiotherapy 2 | From enrolment to analysis, on average 4-6 weeks
  This will involve analysis of radiotherapy plans produced following an MRI scan during radiotherapy treatment and compared to the original radiotherapy plan, to include:
  Volumetric Comparison (assessment of differences in target and OAR delineation volumes);
MRI-Adapted Radiotherapy 3 | From enrolment to analysis, on average 4-6 weeks
  This will involve analysis of radiotherapy plans produced following an MRI scan during radiotherapy treatment and compared to the original radiotherapy plan, to include:
  Prediction of change in toxicity using normal tissue complication probability modelling

OTHER OUTCOMES:
Quantitative Imaging Biomarkers | From enrolment until a maximum of 2 years after completing treatment
  This exploratory end point will involve analysis of the feasibility, sensitivity and specificity of structural and functional MRI sequences identified as potential imaging biomarkers. This will include correlation of the potential imaging biomarker with patient outcomes including histological tumour regression grading for patients who go on to have surgery, disease progression on other radiological imaging (as per RECIST) and with CTCAE toxicity grading following radiotherapy treatment and with survival metrics e.g. progression free survival, cancer specific survival, overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Clair Brunner, MB BChir BA MRCP FRCR PGCert, Principal Investigator — Swansea Bay University Health Board; Jonathan Phillips, PhD MSci MSc PGDip PGCert, Principal Investigator — Swansea Bay University Health Board and Swansea University; Owen Nicholas, MBBS MRCP MD, Principal Investigator — Swansea Bay University Health Board
Locations (1):
- Swansea Bay University Health Board, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keall P, Poulsen P, Booth JT. See, Think, and Act: Real-Time Adaptive Radiotherapy. Semin Radiat Oncol. 2019 Jul;29(3):228-235. doi: 10.1016/j.semradonc.2019.02.005. PMID 31027640
- [Background] Hunt A, Hansen VN, Oelfke U, Nill S, Hafeez S. Adaptive Radiotherapy Enabled by MRI Guidance. Clin Oncol (R Coll Radiol). 2018 Nov;30(11):711-719. doi: 10.1016/j.clon.2018.08.001. Epub 2018 Sep 7. PMID 30201276
- [Background] Bakke KM, Hole KH, Dueland S, Groholt KK, Flatmark K, Ree AH, Seierstad T, Redalen KR. Diffusion-weighted magnetic resonance imaging of rectal cancer: tumour volume and perfusion fraction predict chemoradiotherapy response and survival. Acta Oncol. 2017 Jun;56(6):813-818. doi: 10.1080/0284186X.2017.1287951. Epub 2017 Feb 17. PMID 28464745
- [Background] Huddart R et al, Protocol for Development of daily online magnetic resonance imaging for magnetic resonance image guided radiotherapy, IRAS ID 208449, version 6.0 22/2/2024